CLINICAL TRIAL: NCT01538810
Title: Biomarker Correlates of Radiologic Imaging
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201201061
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Abdominal CT Imaging Performed as Standard of Care
Keywords: CT imaging

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assemble a collection of urine and blood samples for the development and validation of biomarkers potentially useful in correlating or improving the diagnostic utility of abdominal imaging.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Undergoing abdominal CT imaging (standard of care)
* Signed, informed consent

Exclusion Criteria:

* Patients on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anyone undergoing an abdominal image, meeting eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 751 (Actual)
Dates: Start 2012-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Quantitative measures | at enrollment
  Confirm the ability of quantitative measure of AQP-1 and ADFP by ELISA from urine and blood samples to develop and validate an assay for patients with renal cancer.

SECONDARY OUTCOMES:
differentiation of cancerous from non-cancerous renal mass | at analysis
  Correct determination of tumor burden and differentiation of cancerous from non-cancerous renal mass.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Morrissey, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School Of Medicine, St Louis, Missouri, United States